CLINICAL TRIAL: NCT05744479
Title: Metformin for Antipsychotic-induced Weight Gain in Adults With Intellectual Disability: A Double-Blind Randomized Control Trial
Brief Title: Metformin for Antipsychotic-induced Weight Gain in Adults With Intellectual Disability
Acronym: METIDD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 024/2022
Record Dates: First submitted 2023-01-13; First posted 2023-02-27 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2024-08

CONDITIONS: Intellectual Disability; Developmental Disability; Obesity
Keywords: Intellectual Disability; Developmental Disability; Obesity; Metformin
MeSH Terms: conditions — Intellectual Disability; Developmental Disabilities; Obesity | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Metformin vs Placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blinded RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin (Oral) (Experimental): 50 participants will be administered oral metformin titrated to a maximum dose of 2000mg/day for 24 weeks.
  Interventions: Drug: Metformin; Behavioral: Lifestyle Intervention
- Placebo (Placebo Comparator): 50 participants will be administered an identical oral placebo for 24 weeks.
  Interventions: Drug: Placebo; Behavioral: Lifestyle Intervention

INTERVENTIONS:
Drug: Metformin — Metformin oral, 2000mg/day, for 24 weeks.
  Arms: Metformin (Oral)
Drug: Placebo — Oral placebo for 24 weeks
  Arms: Placebo
Behavioral: Lifestyle Intervention — Participants from both groups will meet a dietician and a diabetes educator at the study start to obtain advice regarding healthy diet, portion size, and meal planning to improve physical health. All participants will be invited to monthly group meetings to learn skills which will help them in a variety of wellness areas such as physical exercises and diet. Attendance in these sessions will be encouraged but not mandatory, and attendance will be recorded. Fidelity with these interventions will be captured using diet and physical activity questionnaires at RCT start, midpoint and end, and end of open label phase.

SUMMARY:
People with IDD (intellectual and developmental disability) have very high rates of obesity and die prematurely from cardiometabolic disease. While antipsychotics contribute to this problem, their use is necessary and appropriate in a significant subgroup of individuals with IDD. Exercise and diet interventions have limitations and may not be sufficient, requiring effective adjunctive pharmacological approaches to target obesity and related comorbidities in IDD. However, persons with IDD treated with antipsychotics are systematically excluded from clinical trials hindering development of evidence to help guide safe and effective treatment of these comorbidities. Moreover, evidence from other disorders cannot be extrapolated to IDD given inherent biological differences between disorders. This trial will address the identified gaps, which extend beyond cardiovascular morbidity and negatively impact psychosocial outcomes, in a hugely underserviced population.This is the the first RCT (randomized control trial) to examine the efficacy of metformin in overweight or obese adults with IDD who have experienced antipsychotic-induced weight gain. By generating efficacy data for a very accessible and scalable intervention, allows for guideline and implementation strategies to address a recalcitrant health problem.

ELIGIBILITY:
Inclusion Criteria:

* Stable outpatients
* Age 16-65 years
* Diagnosed with an IDD
* On maintenance treatment with an antipsychotic (stable dose for ≥3 months).
* BMI must be ≥30 kg/m2, OR ≥27 kg/m2 with at least one weight-related comorbidity (treated or untreated) such as: hypertension, dyslipidaemia, obstructive sleep apnea, or impaired fasting glucose, OR >=25 for individuals who have gained > 5% body weight in association with AP use.
* Females of child-bearing age must be on one of the following regular contraceptives:

  1. Agree to abstain from sex for the duration of the trial or
  2. A barrier method of a diaphragm with spermicide and/or Latex condom or
  3. An oral contraceptive agent, implantable contraceptive or an injectable contraceptive for at least six months prior to entering the study and will continue its use throughout the study, or
  4. An intrauterine device, or
  5. Partner has had a vasectomy at least 3 months prior to study start

Exclusion Criteria:

* Females who are nursing, currently pregnant, or have a positive pregnancy test
* Clinical or laboratory evidence of uncompensated cardiovascular, endocrine, haematological, hepatic, renal, or pulmonary disease
* Previous treatment and lack of efficacy or tolerability with metformin
* History or diagnosis of Type 1 Diabetes (T1D) or Type 2 Diabetes (TD2) or fasting blood work, HbA1c > 6.5%
* History of metabolic acidosis or lactic acidosis
* Treatment with weight-lowering agents
* Medications with significant renal impact
* Major medical or surgical event in the preceding 3 months
* Acute suicidal risk.
* Moderate to severe substance use disorder, other than caffein or nicotine use disorder

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Individual's percentage change in body weight | Weeks 0, 4, 8, 12, 16, 10, 24
  Percentage change in body weight measured in percentage change of pounds (lbs)

SECONDARY OUTCOMES:
Proportion of participants who achieve body weight reduction ≥5%, and ≥10% in each arm | Week 0 and week 24
  Percentage change in body weight measured in percentage change of pounds (lbs), expressed as a percentage
Between group (metformin vs placebo) absolute change in weight | Week 24
  Absolute change in body weight between metformin and placebo groups measured in pounds (lbs). Calculated by the mean change in weight between the metformin and placebo groups.
Between group absolute change in waist circumference | Week 24
  Absolute change in waist circumstance measured in centimetres (cm) between metformin and placebo groups. Calculated by the mean change in waist circumstance between the metformin and placebo groups.
Between group absolute change in BMI | Week 24
  Absolute change in BMI between metformin and placebo groups. Calculated by the mean change in BMI between the metformin and placebo groups.
Change in whole body insulin sensitivity calculated with Matsuda Index | Week 0 and Week 24
  With the results of the oral glucose tolerance test at Week 0 and Week 24, insulin sensitivity was calculated with the Matsuda index.
  Insulin sensitivity was calculated with Matsuda index: [10,000 / √glucose minute 0 x insulin minute 0) (mean glucose (OGTT) x mean insulin OGTT)]. A higher result is better.
  In the formula OGTT: oral glucose tolerance test.
Change in beta-cell function, measured using the Insulin Secretion-Sensitivity Index-2 (ISSI-2) | Week 0 and Week 24
  ISSI-2 is defined as the product of (i) insulin secretion measured by the ratio of the area-under-the-insulin-curve to the area-under-the-glucose curve and (ii) insulin sensitivity measured by the Matsuda index.
Proportion in each group converting to impaired glucose tolerance, prediabetes, or type 2 diabetes | Week 0 and Week 24
  Measured through the change in HOMA-IR (Homeostatic Model Assessment for Insulin Resistance) derived from the Oral Glucose Tolerance Test (OGTT).
Change in cardiovascular risk factors assessed by change in C-reactive protein | Week 0 and Week 24
  Measured through the change in C-reactive protein (CRP) assessed at week 0 and week 24.
  Healthy levels:
  CRP: Less than 0.3 mg/dL
Change in cardiovascular risk factor assessed by change in fasting lipids profile | Week 0 and Week 24
  Change in fasting lipid profile (low-density lipoprotein cholesterol (LDL), high-density lipoprotein cholesterol (HDL), and triglycerides) assessed at week 0 and week 24.
  Healthy levels:
  LDL: less than 100mg/dL HDL: 40mg/dL or higher Triglycerides: less than 150mg/dL
Change in cardiovascular risk factor assessed by change in blood pressure | Week 0 and Week 24
  Measured through the change in blood pressure (systolic/diastolic) assessed at week 0 and week 24. A blood pressure range of 110/70 to 120/80 is considered normal.
Change in visceral and liver fat content | Week 0 and Week 24
  Change in visceral and liver fat content assessed via MRI scans at week 0 and week 24.
Medication Adherence | Week 0 to Week 24
  Measured through returning of blister pill packs, and assessing number of pills taken.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada